CLINICAL TRIAL: NCT03727048
Title: Effect of Toradol on Post-operative Foot and Ankle Healing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Principal Investigator, Tiffany Morrison, MS, Director of Clinical Trials, Rothman Institute Orthopaedics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016Raikin
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Ankle Fractures; Trauma Injury
MeSH Terms: conditions — Ankle Fractures; Accidental Injuries | interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): To the control group post ankle fracture surgery, per subject 30 tablets of 5/325 oxycodone-acetaminophen with instructions to take 1 or 2 tabs every 4 to 6 hours as needed for pain
  Interventions: Other: No ketorolac
- Intervention (Experimental): To the treatment group post ankle fracture surgery, per subject 30mg of IV ketorolac intraoperatively; 20 tablets of 10mg ketorolac with instructions to take every 6 hours, and 30 tablets of 5/325 oxycodone-acetaminophen with instructions to take 1 or 2 tabs every 4 to 6 hours as needed for pain
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — the investigators aimed to evaluate the effect of postoperative ketorolac after ankle fracture surgery on postoperative opioid consumption, pain control, an patient satisfaction.
  Other Names: Toradol
  Arms: Intervention
Other: No ketorolac — standard of care post operative pain management protocol
  Arms: Control

SUMMARY:
The use of Toradol for pain control in surgical orthopedic cases is currently a topic of interest within the field. The proposed study is a prospective randomized study evaluating postoperative pain, opioid requirement, complication/reoperation rates and nonunion rates in patients undergoing surgical treatment for isolated lateral malleolar fibula fractures. Patients will be randomized to either the Treatment Group (Toradol) or the Control Group (Non-Toradol). Both Toradol and non-Toradol drug regimens are currently prescribed by the Foot and Ankle Team at the Rothman Institute and this study will serve as a valuable comparison.

ELIGIBILITY:
Inclusion Criteria:

* patients over age of 18 undergoing outpatient open reduction and internal fixation (ORIF) by a fellowship-trained foot and ankle orthopaedic surgeon for isolated lateral malleolar, bimalleolar, or trimalleolar ankle fractures.

Exclusion Criteria:

* open fracture
* allergies to one or more of the study medications
* existing use of narcotics
* renal insufficiency as defined by history and preoperative creatinine level
* pregnancy
* hospital admittance

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2016-08; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Visual analog score for pain | Days 1-7 post-op
  To evaluate the pain VAS scores of all patients

SECONDARY OUTCOMES:
Opioid pill intake | Days 1-7 post-op
  opioid requirement
Radiographic healing | 12-33 weeks
  Ankle fracture healing post op via radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Steven Raikin, MD, Principal Investigator — Rothman Orthopaedic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cappello T, Nuelle JA, Katsantonis N, Nauer RK, Lauing KL, Jagodzinski JE, Callaci JJ. Ketorolac administration does not delay early fracture healing in a juvenile rat model: a pilot study. J Pediatr Orthop. 2013 Jun;33(4):415-21. doi: 10.1097/BPO.0b013e318288b46f. PMID 23653032
- [Background] Jeffcoach DR, Sams VG, Lawson CM, Enderson BL, Smith ST, Kline H, Barlow PB, Wylie DR, Krumenacker LA, McMillen JC, Pyda J, Daley BJ; University of Tennessee Medical Center, Department of Surgery. Nonsteroidal anti-inflammatory drugs' impact on nonunion and infection rates in long-bone fractures. J Trauma Acute Care Surg. 2014 Mar;76(3):779-83. doi: 10.1097/TA.0b013e3182aafe0d. PMID 24553548
- [Background] Reikeraas O, Engebretsen L. Effects of ketoralac tromethamine and indomethacin on primary and secondary bone healing. An experimental study in rats. Arch Orthop Trauma Surg. 1998;118(1-2):50-2. doi: 10.1007/s004020050310. PMID 9833106
- [Background] Glassman SD, Rose SM, Dimar JR, Puno RM, Campbell MJ, Johnson JR. The effect of postoperative nonsteroidal anti-inflammatory drug administration on spinal fusion. Spine (Phila Pa 1976). 1998 Apr 1;23(7):834-8. doi: 10.1097/00007632-199804010-00020. PMID 9563116
- [Background] Li Q, Zhang Z, Cai Z. High-dose ketorolac affects adult spinal fusion: a meta-analysis of the effect of perioperative nonsteroidal anti-inflammatory drugs on spinal fusion. Spine (Phila Pa 1976). 2011 Apr 1;36(7):E461-8. doi: 10.1097/BRS.0b013e3181dfd163. PMID 20489674
- [Background] Reuben SS, Ablett D, Kaye R. High dose nonsteroidal anti-inflammatory drugs compromise spinal fusion. Can J Anaesth. 2005 May;52(5):506-12. doi: 10.1007/BF03016531. PMID 15872130
- [Background] Pradhan BB, Tatsumi RL, Gallina J, Kuhns CA, Wang JC, Dawson EG. Ketorolac and spinal fusion: does the perioperative use of ketorolac really inhibit spinal fusion? Spine (Phila Pa 1976). 2008 Sep 1;33(19):2079-82. doi: 10.1097/BRS.0b013e31818396f4. PMID 18698276
- [Background] McDonald E, Winters B, Nicholson K, Shakked R, Raikin S, Pedowitz DI, Daniel JN. Effect of Postoperative Ketorolac Administration on Bone Healing in Ankle Fracture Surgery. Foot Ankle Int. 2018 Oct;39(10):1135-1140. doi: 10.1177/1071100718782489. Epub 2018 Jul 4. PMID 29972028
- [Background] Donohue D, Sanders D, Serrano-Riera R, Jordan C, Gaskins R, Sanders R, Sagi HC. Ketorolac Administered in the Recovery Room for Acute Pain Management Does Not Affect Healing Rates of Femoral and Tibial Fractures. J Orthop Trauma. 2016 Sep;30(9):479-82. doi: 10.1097/BOT.0000000000000620. PMID 27124828